CLINICAL TRIAL: NCT03939689
Title: A Multicenter, Randomized, Controlled Phase 2 Study: Efficacy and Safety of I-131-1095 Radiotherapy in Combination With Enzalutamide in mCRPC Patients Who Are 18F-DCFPyL PSMA-avid, Chemotherapy-naïve, and Progressed on Abiraterone (ARROW )
Brief Title: I-131-1095 Radioligand Plus Enzalutamide vs Enzalutamide for mCRPC That Progressed During Abiraterone (ARROW).
Acronym: ARROW
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1095-2301
Record Dates: First submitted 2019-05-03; First posted 2019-05-07 (Actual); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Prostate Cancer; Castration-resistant Prostate Cancer; Prostatic Neoplasm; Cancer of the Prostate; Progressive mCRPC
Keywords: bone metastases; 18F-DCFPyL; PSMA PET; PSMA-avidity; biomarker; radioligand therapy; adjunct radiation therapy; dosimetry; SPECT/CT; docetaxel
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Intervention Model Description: The study population includes patients with PSMA-avid mCRPC whose disease has progressed despite abiraterone therapy, and are planned for treatment with enzalutamide.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Enzalutamide (Active Comparator): Participants received the label dosage of enzalutamide once daily for up to 53 weeks.
  Interventions: Drug: Enzalutamide
- I-131-1095 in combination with enzalutamide (Experimental): Participants received up to 4 (8-week) cycles of I-131-1095: 100 mCi for the first dose. Subsequent dose(s) were reduced to 75 mCi for participants experiencing any of the dose-limiting toxicities. The third and fourth therapeutic doses could be reduced to 75 mCi on the basis of dosimetry assessment after administration of 10 mCi of I-131-1095 prior to the third dosing cycle. Participants also received the label dosage of enzalutamide once daily for up to 53 weeks.
  Interventions: Drug: I-131-1095; Drug: Enzalutamide

INTERVENTIONS:
Drug: I-131-1095 — Participants received up to 4 (8-week) cycles of I-131-1095: 100 mCi for the first dose. Subsequent dose(s) were reduced to 75 mCi for participants experiencing any dose-limiting toxicities. The third and fourth therapeutic doses could be reduced to 75 mCi on the basis of dosimetry assessment after administration of 10 mCi of I-131-1095 prior to the third dosing cycle. Participants also received the label dosage of enzalutamide once daily for up to 53 weeks.
  Other Names: 131 I-PSMA-1095; 131I-LNTH-1095
  Arms: I-131-1095 in combination with enzalutamide
Drug: Enzalutamide — Participants received the label dosage of enzalutamide once daily for up to 53 weeks.
  Other Names: Xtandi

SUMMARY:
This clinical trial was done to show whether a radioactive drug (I-131-1095) that binds to prostate-specific membrane antigen (PSMA) is useful in treating metastatic prostate cancer that is positive for PSMA. The trial enrolled men whose PSMA-positive metastatic prostate cancer had progressed while they were taking abiraterone. During the trial, all of the men took enzalutamide (standard-of-care therapy) once a day. However, some of the men also had up to 4 doses (8 weeks apart) of I-131-1095 (in addition to taking enzalutamide once a day). At specified times during the trial, all of the men had blood tests (to measure levels of prostate-specific antigen [PSA]) and imaging studies (to assess tumor status). The two groups of men were then compared in several ways. The main comparison was the percentage of men in each group with at least a 50% decrease in PSA levels. Other comparisons involved the response of the tumors (as seen on imaging) and overall survival. To assess safety, the number of adverse events in both groups were also compared.

DETAILED DESCRIPTION:
This phase 2 clinical trial (conducted in the United States and Canada) enrolled chemotherapy-naïve men whose PSMA-positive (as shown by piflufolastat F18 imaging) metastatic prostate cancer had progressed during treatment with abiraterone. The participants were stratified by risk factors at Screening and then randomized 2:1 either to receive PSMA radioligand therapy (up to four 8-week cycles of I-131-1095) plus standard treatment with enzalutamide or to receive standard treatment with enzalutamide as monotherapy. The prostate-specific antigen (PSA) levels and radiographic response or progression (RECIST v1.1 criteria for soft tissue and PCWG3 criteria for bone) were then monitored for up to 53 weeks of randomized treatment. The primary outcome measure was PSA response rate (percentage of participants with a confirmed ≥50% decrease in serum PSA). Other outcome measures included percentage of participants with partial or complete response (radiographic), duration of response, time to progression (PSA or radiographic), time to next treatment for prostate cancer, and overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Male ≥ 18 years of age
2. Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features at initial diagnosis
3. Castration-resistant prostate cancer, with serum testosterone ≤ 50 ng/dL at Screening
4. Radiographic evidence of metastatic disease prior to Randomization or up to 21 days prior to Screening
5. Disease progression on prior abiraterone therapy as defined by meeting at least one of the following criteria per the investigator:

   1. PSA progression as defined by a minimum of two rising PSA levels at least 1 week apart
   2. Soft tissue disease progression defined by RECIST 1.1
   3. Bone disease progression defined by two or more new lesions on bone scan
6. Planned to receive treatment with enzalutamide
7. Subjects who are ineligible or choose not to receive taxane-based chemotherapy based on personal preference or physician opinion. Examples of conditions that could make a patient ineligible or refuse to receive taxane-based chemotherapy, but would allow them to still be eligible to receive I-131-1095 include the following:

   1. Poor performance status
   2. Prior intolerance to cytotoxic agents
   3. History of another malignancy suspected for recurrence or metastases
   4. Other serious medical conditions such as symptomatic peripheral neuropathy CTCAE Grade 2 or higher; or clinically significant cardiovascular disease per the Investigator or treating physician
8. Subjects receiving bisphosphonate therapy must have been on stable doses for at least 4 weeks prior to Randomization
9. ECOG performance status 0-2
10. If sexually active, agree to use a medically acceptable method of birth control or sexual abstinence from the time of dosing through 28 days after the last dose of I-131-1095. Female partners must use hormonal or barrier contraception unless postmenopausal or abstinent.
11. Estimated life expectancy of at least 6 months as determined by the Investigator.
12. Able and willing to provide signed informed consent and comply with protocol requirements

Exclusion Criteria:

1. Received any anti-tumor therapy within 4 weeks of Randomization, with the exception of abiraterone, GnRH therapy and non-radioactive bone-targeted agents
2. Received prior chemotherapy for castration-resistant prostate cancer
3. Superscan as evidenced on baseline bone scan
4. Treatment with Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Radium-223 within 6 months prior to Randomization
5. Prior hemi-body irradiation
6. Prior PSMA-targeted radioligand therapy
7. Major surgery within 4 weeks of Randomization
8. Impaired organ function as evidenced by the following laboratory values at Screening:

   1. Absolute neutrophil count < 1500 μL
   2. Platelet count < 100,000/μL
   3. Hemoglobin < 9.5 g/dL
   4. Albumin < 3.0 g/dL (30 g/L)
   5. Total bilirubin > 2 x ULN unless in instances of known or suspected Gilbert's disease
   6. AST or ALT > 2.5 x ULN
   7. Calculated creatinine clearance (CrCL) < 30 mL/min (Cockroft-Gault equation), or currently on renal dialysis.
9. QT interval corrected for heart rate (QTc) > 470 msec
10. Previous use of enzalutamide for more than 7 days prior to consent
11. Planned initiation of alternative therapy for prostate cancer, investigational therapy, or participation in clinical trials during the study
12. History or risk of seizure (i.e., clinically significant neurological disorder) or any other condition that contraindicates treatment with enzalutamide
13. Gastrointestinal disorder affecting absorption of oral medications
14. Known or suspected brain metastasis or active leptomeningeal disease
15. Active malignancy other than prostate cancer, with the exception of curatively treated non-melanoma skin cancer, carcinoma in situ, or non-muscle invasive bladder/urothelial cancer
16. Subjects with any medical condition or other circumstances that, in the opinion of the investigator, compromise obtaining reliable data, achieving study objectives, or completing the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2024-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Provost, MD, Study Director — Progenics Pharmaceuticals, Inc.
Locations (27):
- United States (20):
  - City of Hope, Duarte, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - UCLA, Los Angeles, California
  - Hoag Family Cancer Institute, Newport Beach, California
  - VA Palo Alto Healthcare System, Palo Alto, California
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - The University of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Tulane Medical School, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - SUNY Upstate Medical University, Syracuse, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - LifeSpan Cancer Institute, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Washington - Seattle Cancer Care Alliance, Seattle, Washington
- Canada (7):
  - The Ottawa Hospital, Ottawa, Ontario
  - London Health Sciences Centre, Toronto, Ontario
  - University Health Network - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre Hospitalier Del' Universite de Montreal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Afshar-Oromieh A, Haberkorn U, Zechmann C, Armor T, Mier W, Spohn F, Debus N, Holland-Letz T, Babich J, Kratochwil C. Repeated PSMA-targeting radioligand therapy of metastatic prostate cancer with 131I-MIP-1095. Eur J Nucl Med Mol Imaging. 2017 Jun;44(6):950-959. doi: 10.1007/s00259-017-3665-9. Epub 2017 Mar 9. PMID 28280855
- [Background] Zechmann CM, Afshar-Oromieh A, Armor T, Stubbs JB, Mier W, Hadaschik B, Joyal J, Kopka K, Debus J, Babich JW, Haberkorn U. Radiation dosimetry and first therapy results with a (124)I/ (131)I-labeled small molecule (MIP-1095) targeting PSMA for prostate cancer therapy. Eur J Nucl Med Mol Imaging. 2014 Jul;41(7):1280-92. doi: 10.1007/s00259-014-2713-y. Epub 2014 Feb 28. PMID 24577951

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by physician referral at academic medical centers in the United States and Canada. Of 28 sites activated, 23 sites (16 in the United States and 7 in Canada) enrolled at least 1 participant. The study was initiated on 30May2019. The first participant consented on 07Jun2019 and last participant consented on 10Jun2022.
Pre-assignment Details: A total of 177 participants were screened.
  Of 132 participants who underwent piflufolastat imaging, 123 met the inclusion criterion of PSMA avidity.
Groups:
- Enzalutamide: Enzalutamide: Enzalutamide will be given orally once daily as prescribed by the physician as standard of care.
- I-131-1095 in Combination With Enzalutamide: I-131-1095: I-131-1095 will be administered intravenously at 100 mCi for the initial therapeutic dose, and up to 3 additional dose(s) at 75 mCi or 100 mCi each, administered at least 8 weeks apart as determined by dosimetry evaluation and occurrence of dose-limiting events.
  Enzalutamide: Enzalutamide will be given orally once daily as prescribed by the physician as standard of care.
Period: Overall Study
Arm/Group | Enzalutamide | I-131-1095 in Combination With Enzalutamide
Started | 39 | 76
Completed | 13 | 29
Not Completed | 26 | 47
Not completed — Radiographic progression | 14 | 17
Not completed — Treatment is no longer benefiting participant | 5 | 6
Not completed — Adverse Event | 1 | 8
Not completed — Unequivocal clinical progression | 2 | 5
Not completed — Other | 1 | 4
Not completed — Death | 0 | 3
Not completed — Participant decision | 0 | 3
Not completed — Withdrawal of consent | 2 | 1
Not completed — Investigator decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: One subject who had not undergone the required PSMA imaging at Screening was randomized. Two of the randomized subjects were later found to be screen failures.
Groups:
- Enzalutamide: Participants received the labeled dosage of enzalutamide once daily for up to 53 weeks.
- Total: Total of all reporting groups
Arm/Group | Enzalutamide | I-131-1095 in Combination With Enzalutamide | Total
Number analyzed (Participants) | 39 | 76 | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 19 | 30
  >=65 years | 28 | 57 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (8.97) | 70.9 (8.96) | 70.7 (8.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 39 | 76 | 115
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 36 | 71 | 107
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 31 | 64 | 95
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 4 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 45 | 74
  Canada | 10 | 31 | 41
Height [Mean (Standard Deviation); unit: cm] | 174.3 (6.52) | 174.7 (7.53) | 174.6 (7.18)
Weight [Mean (Standard Deviation); unit: kg] | 90.77 (18.280) | 90.58 (17.467) | 90.64 (18.008)
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 29.73 (5.350) | 29.66 (4.629) | 29.68 (4.861)

OUTCOME MEASURES:

1. Primary Outcome: PSA Response Rate
Description: The percentage of participants with a PSA response according to PCWG3 criteria. PCWG3 defines PSA response as the first occurrence of a 50 percent or more decline in PSA from baseline, confirmed by a second measurement at least 3 weeks later.
Time Frame: Up to 53 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide | I-131-1095 in Combination With Enzalutamide
Number analyzed (Participants) | 39 | 76
Participants | 10 | 44
Statistical Analysis 1: Comparison: Enzalutamide vs I-131-1095 in Combination With Enzalutamide; A Cochran-Mantel-Haenszel (CMH) test with adjustment for stratification factor (prostate cancer risk factor at Screening) was carried out by using complete cases for the FAS population (missing data were not imputed for this analysis). Intermediate risk at Screening: hemoglobin (Hgb) ≥11 g/dL and LDH <262 IU/L and ALP <414 IU/L. High-risk at Screening: Hgb <11 g/dL or LDH ≥262 IU/L or ALP ≥414 IU/L; Test type: Superiority; p = 0.0025, Cochran-Mantel-Haenszel

2. Secondary Outcome: Objective Response Rate (ORR)
Description: The proportion of participants who have a partial response (PR) or complete response (CR) based on RECIST 1.1 for soft tissue or PCWG3 for bone (PCWG3-modified RECIST 1.1).
Time Frame: Up to 53 weeks
Measure: Count of Participants; unit: Participants
Groups:
- I-131-1095 in Combination With Enzalutamide: Participants received up to 4 (8-week) cycles of I-131-1095: 100 mCi for the first dose. Subsequent dose(s) reduced to 75 mCi for participants experiencing any of the dose-limiting toxicities. The third and fourth therapeutic doses could be reduced to 75 mCi on the basis of dosimetry assessment after administration of 10 mCi of I-131-1095 prior to the third dosing cycle. Participants also received the label dosage of enzalutamide once daily for up to 53 weeks.
Arm/Group | Enzalutamide | I-131-1095 in Combination With Enzalutamide
Number analyzed (Participants) | 39 | 76
Participants | 4 | 7
Statistical Analysis 1: Comparison: Enzalutamide vs I-131-1095 in Combination With Enzalutamide; Test type: Superiority; p = 0.8060, Chi-squared — The p-value is based on the chi-squared test of the difference in proportions between treatment groups if expected cell frequencies are all greater than 5; otherwise, the p-value is from the Fisher's exact test

3. Secondary Outcome: Radiographic Progression Free Survival (rPFS)
Description: Time from randomization to the first occurrence of radiographic progression based on RECIST 1.1 for soft tissue (≥20% increase in the sum of the longest diameter of the target lesions [relative to the smallest value recorded since the treatment started] or the appearance of ≥1 new lesion) or PCWG3-modified RECIST 1.1 for bone, respectively, or unequivocal clinical progression, or death on study from any cause.
Time Frame: Up to 5 years.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide | I-131-1095 in Combination With Enzalutamide
Number analyzed (Participants) | 39 | 76
Months | 11.5 [2.79 to 18.43] | 14.0 [8.64 to 18.20]
Statistical Analysis 1: Comparison: Enzalutamide vs I-131-1095 in Combination With Enzalutamide; Kaplan-Meier analysis and Greenwood formula used for estimating event-free rates and 95% confidence intervals; Test type: Superiority; p = .5924, Log Rank — Log-rank test of no difference between treatment groups, stratified by prostate cancer risk groups

4. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival is defined as time from randomization to death from any cause.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide | I-131-1095 in Combination With Enzalutamide
Number analyzed (Participants) | 39 | 76
Months | 22.0 [14.59 to NA] — The upper limit of the 95% confidence interval could not be calculated because too few participants had reached the endpoint. | 18.8 [15.34 to 29.47]
Statistical Analysis 1: Comparison: Enzalutamide vs I-131-1095 in Combination With Enzalutamide; Kaplan-Meier analysis and Greenwood formula used for estimating event-free rates and 95% confidence intervals; Test type: Superiority; p = 0.5924, Log Rank — Log-rank test of no difference between treatment groups, stratified by prostate cancer risk groups

5. Secondary Outcome: PSA Progression
Description: Time from randomization to the date of the first PSA increase from baseline ≥ 25 percent and ≥ 2 ng/ml above nadir confirmed by a second PSA assessment defining progression ≥ 3 weeks later per PCWG3.
Time Frame: Up to 53 weeks
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide | I-131-1095 in Combination With Enzalutamide
Number analyzed (Participants) | 39 | 76
Months | 10 [3.45 to NA] — The upper limit of the 95% confidence interval could not be calculated because not enough participants had reached the endpoint. | NA [6.97 to NA] — The median cannot be calculated until at least 50% of the participants have reached the endpoint. The upper limit of the 95% confidence interval could not be calculated because not enough participants had reached the endpoint.
Statistical Analysis 1: Comparison: Enzalutamide vs I-131-1095 in Combination With Enzalutamide; Event-free rates and 95% CI were estimated by using Kaplan-Meier method and Greenwood formula; Test type: Superiority; p = 0.6199, Log Rank — P value from the log-rank test of no difference between treatment groups, stratified by prostate cancer risk group at Screening

6. Secondary Outcome: Duration of Response
Description: Time from the first date of complete response (CR) or partial response (PR) to the first occurrence of radiographic progression based on PCWG3-modified RECIST 1.1, or unequivocal clinical progression. Complete response was defined as disappearance of all target lesions. Partial response was defined as ≥30% decrease from baseline in the sum of the longest diameter of target lesions.
Time Frame: Up to 5 years.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide | I-131-1095 in Combination With Enzalutamide
Number analyzed (Participants) | 39 | 76
Months | 15.1 [3.29 to NA] — The upper limit of the 95% confidence interval could not be calculated because not enough participants had reached the endpoint | 15.0 [3.29 to NA] — The upper limit of the 95% confidence interval could not be calculated because not enough participants had reached the endpoint.
Statistical Analysis 1: Comparison: Enzalutamide vs I-131-1095 in Combination With Enzalutamide; Event free rates and 95% CI were estimated by using Kaplan-Meier method and Greenwood formula; Test type: Superiority; p = .1823, Log Rank — P-value from the log-rank test of no difference between treatment groups, stratified by prostate cancer risk group at Screening

7. Secondary Outcome: Time to Initiation of Next Treatment for Prostate Cancer
Description: Time from randomization to initiation of any new treatment for prostate cancer.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: Time to event, months
Arm/Group | Enzalutamide | I-131-1095 in Combination With Enzalutamide
Number analyzed (Participants) | 39 | 76
Time to event, months | 10.9 [5.16 to 13.60] | 18.3 [13.14 to NA] — The upper limit of the 95% confidence interval could not be calculated because not enough participants had reached the endpoint.
Statistical Analysis 1: Comparison: Enzalutamide vs I-131-1095 in Combination With Enzalutamide; Event-free rates and 95% CI were estimated by using Kaplan-Meier method and Greenwood formula; Test type: Superiority; p = 0.0006, Log Rank — [p-value comment as in outcome 6, analysis 1]

ADVERSE EVENTS:
Time Frame: Randomized treatment phase (up to 53 weeks)
Description: Adverse events were recorded during the randomized treatment phase (up to 53 weeks). Participants were also followed for clinical progression or death for up to 5 years after start of treatment.
Arm/Group | Enzalutamide | I-131-1095 in Combination With Enzalutamide
All-Cause Mortality (participants affected / at risk) | 1/39 | 3/76
Serious Adverse Events (participants affected / at risk) | 11/39 | 29/76
Other Adverse Events (participants affected / at risk) | 37/39 | 72/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enzalutamide (N=39) | I-131-1095 in Combination With Enzalutamide (N=76)
Anemia (Blood and lymphatic system disorders) | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 2
Platelet count decreased/Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Aplastic anaemia (Blood and lymphatic system disorders) | 0 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
White blood cell count decreased/Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Fatigue/Asthenia (General disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 2
Abdominal infection (Gastrointestinal disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Groin abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Subdural hematoma (Injury, poisoning and procedural complications) | 0 | 1
Platelet count decreased/Thrombocytopenia (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Spinal cord compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Haematuria (Renal and urinary disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Enzalutamide (N=39) | I-131-1095 in Combination With Enzalutamide (N=76)
Fatigue (General disorders) | 20 | 54
Nausea (Gastrointestinal disorders) | 12 | 44
Decreased appetite (Metabolism and nutrition disorders) | 7 | 36
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 23
Dry mouth (Gastrointestinal disorders) | 1 | 36
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 23
Anaemia (Blood and lymphatic system disorders) | 6 | 27
Diarrhoea (Gastrointestinal disorders) | 9 | 18
Weight decreased (Immune system disorders) | 6 | 20
Vomiting (Gastrointestinal disorders) | 6 | 19
Platelet count decreased (Blood and lymphatic system disorders) | 0 | 23
Headache (Nervous system disorders) | 6 | 15
Dysgeusia (Nervous system disorders) | 2 | 17
Constipation (Gastrointestinal disorders) | 5 | 13
Lymphocyte count decreased (Blood and lymphatic system disorders) | 2 | 15
Dizziness (Nervous system disorders) | 4 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 15
Oedema peripheral (General disorders) | 3 | 11
Hypothyroidism (Endocrine disorders) | 0 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 8
Insomnia (Psychiatric disorders) | 4 | 7
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 | 4
Blood thyroid stimulating hormone increased (Investigations) | 0 | 9
Fall (Injury, poisoning and procedural complications) | 3 | 6
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 | 8
Haematuria (Renal and urinary disorders) | 2 | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 5
Rash (Skin and subcutaneous tissue disorders) | 3 | 5
White blood cell count decreased (Blood and lymphatic system disorders) | 1 | 7
Chills (General disorders) | 1 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Hot flush (Vascular disorders) | 4 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 7
Neutropenia (Blood and lymphatic system disorders) | 0 | 7
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 6
Contusion (Injury, poisoning and procedural complications) | 0 | 6
Paraesthesia (Nervous system disorders) | 2 | 4
Anxiety (Psychiatric disorders) | 1 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Hypertension (Vascular disorders) | 2 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 4
Pyrexia (General disorders) | 0 | 5
Urinary tract infection (Infections and infestations) | 1 | 4
Amnesia (Nervous system disorders) | 0 | 4
Depression (Psychiatric disorders) | 2 | 2
Dry eye (Eye disorders) | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 4
Haemoglobin decreased (Investigations) | 0 | 4
Pain (General disorders) | 0 | 4
Pancytopenia (Blood and lymphatic system disorders) | 0 | 4
Taste disorder (Nervous system disorders) | 0 | 4
Cardiac murmur (Investigations) | 2 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 1
Malaise (General disorders) | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1
Non-cardiac chest pain (General disorders) | 3 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 | 0
Swollen tongue (Gastrointestinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/89/NCT03939689/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-03): https://cdn.clinicaltrials.gov/large-docs/89/NCT03939689/SAP_001.pdf